CLINICAL TRIAL: NCT05464680
Title: Pulmonary Diffusion of Antibiotics During Mechanically Ventilated Pneumonia in Patients Admitted for ARDS Following SARS-CoV-2 Pneumonia
Brief Title: Pulmonary Diffusion of Antibiotics in Patients Admitted for ARDS Following SARS-CoV-2 Pneumonia
Acronym: ATB-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM21_0415; ID-RCB (Other: 2021-A03122-39)
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: ARDS; SARS-CoV 2 Pneumonia
Keywords: mechanical ventilation; antibiotics diffusion; ARDS; SARS-CoV 2
MeSH Terms: interventions — Blood Specimen Collection; Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients positive to SARS-CoV 2 (Experimental): Patients admitted to the ICU and placed on VM following SARS-CoV-2 pneumonia
  Interventions: Other: blood sample and bronchoalveolar lavage
- Patients negative to SARS-CoV 2 (Sham Comparator): Patients admitted to the ICU and placed on VM outside of SARS-CoV-2 pneumonia
  Interventions: Other: blood sample and bronchoalveolar lavage

INTERVENTIONS:
Other: blood sample and bronchoalveolar lavage — These patients are put on VM as part of their care and present a suspicion of a 1st episode of PAVM for which a microbiological sample is taken and a probabilistic antibiotic therapy is started with the PIP-TAZ association (D0). A plasma PIP-TAZ assay will be performed 48 hours after the start of antibiotic therapy with PIP-TAZ. Blood urea will be measured and a mini-LBA (performed with a Combicatheter®) will be performed to measure PIP-TAZ and urea in the ELF.
  On day 7 of the antibiotic therapy (last day of the planned antibiotic therapy), the same samples are taken and the same analyses are performed + bacteriology on the mini BAL. For patients for whom antibiotic therapy has been interrupted because of sterile samples, the samples taken at D7 will not be taken.
  The clinical outcome of the patient will then be recorded until D60.

SUMMARY:
Patients on mechanical ventilation (MV) following SARS-CoV-2 pneumonia frequently develop ventilator-associated pneumonia (VAP). The incidence of MVAP during SARS-CoV-2 infections ranges from 50 to nearly 90%. In addition, up to 80% of recurrences of VAP (a new episode, most often attributable to the same bacteria) have been described, reflecting the failure of the initial antibiotic therapy. This incidence is much higher than that described for other etiologies of acute respiratory distress syndrome (ARDS). The investigators hypothesize that during VAP, there is an alteration of the diffusion of intravenous antibiotics in the lung parenchyma in COVID-19 patients in relation to several factors characteristic of SARS-CoV-2 infection. This altered diffusion may explain the high number of recurrences of MVAP compared to non-COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient over 18 years of age 2. Patient has given consent or consent obtained from the trusted person if the patient is not capable of consenting, after informed consent.

  3. Patient with ARDS 4. Patient requiring MV for ARDS (as defined by Berlin (15)), regardless of etiology (COVID-19 or other cause of ARDS) 5. Patient with suspected 1st episode of ARDS for which microbiological sampling is performed (bronchial aspiration, protected distal sampling (PDS), bronchoalveolar lavage (BAL)) 6. Patients who have received probabilistic antibiotic therapy within 24 hours of the microbiological sample, including piperacillin-tazobactam (PIP-TAZ) administered according to current recommendations.

  7. Patient who is a beneficiary of or affiliated to a social security system

Exclusion Criteria:

1. Patients for whom PIP-TAZ is administered as a discontinuous infusion.
2. Contraindication to the realization of a mini-LBA: patient whose respiratory state is too precarious for the realization of a mini-LBA for intra pulmonary antibiotics dosage (SpO2<94% under FiO2 100% under VM), presence of a non drained pneumothorax, bronchial prosthesis, recent bronchial suture
3. Patient with a second episode of PAVM.
4. Patients with KDIGO stage ≥ 3 renal failure or extra-renal replacement therapy (creatinine measurement on the day of inclusion, performed as part of routine care).
5. Patient on ExtraCorporeal Membrane Oxygenation (ECMO) or ExtraCorporeal CO2 Removal (ECCO2R).
6. Pregnant or breastfeeding women, patients under guardianship or trusteeship, deprived of liberty
7. Patients who are moribund or for whom limitations of active therapies have been decided.
8. Any condition, which in the opinion of the investigator, would not allow the implementation of the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Compare the pulmonary diffusion of piperacillin | 48 hours following antibiotics administration
  Dosage in the epithelial lining fluid

SECONDARY OUTCOMES:
Pulmonary diffusion of tazobactam | 48 hours following antibiotics administration
  Dosage in the epithelial lining fluid
Concentrations of piperacillin in effective pulmonary and plasma targets | 48 hours following antibiotics administration
  Piperacillin concentrations in Epithelial Lining Fluid
Concentrations of piperacillin in effective pulmonary and plasma targets | 7 days following antibiotics administration
  Piperacillin concentrations in plasma
Concentrations of tazobactam in effective pulmonary and plasma targets | 7 days following antibiotics administration
  Tazobactam concentrations in Epithelial Lining Fluid
Concentrations of tazobactam in effective pulmonary and plasma targets | 48 hours following antibiotics administration
  Tazobactam concentrations in Epitehlial Lining Fluid and plasma separately at H48 and 7 days after initiation of antibiotic therapy

CONTACTS AND LOCATIONS:
Overall Officials: François Cremieux, Study Director — AP-HM
Locations (1):
- Service Médecine Intensive Réanimation, Marseille, France

IPD SHARING:
Plan to Share IPD: No